CLINICAL TRIAL: NCT01216852
Title: A Single Dose, 2-Period, 2-Treatment Bioequivalency Study of Losartan Potassium Tablets 100 mg Under Fasted Conditions
Brief Title: Bioequivalency Study of Losartan Potassium 100 mg Tablet Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director - Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LOSA-01
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Losartan Potassium — 100 mg tablet
  Other Names: COZAAR

SUMMARY:
The objective of this study was to prove the bioequivalence of Losartan Potassium 100 tablet under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to losartan potassium or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-08; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis N. Morrison, D.O., Principal Investigator — Bio-Kinetic Clinical Applications, Inc.
Locations (1):
- Bio-Kinetic Clinical Applications, Inc., Springfield, Missouri, United States